CLINICAL TRIAL: NCT01291017
Title: A Phase II Clinical Trail of the Cyclin Dependent Kinase (CDK)4/6 Inhibitor, PD0332991 in Previously Treated, Advanced NSCLC Patients With Wildtype Retinoblastoma Protein (RB) and Inactive Cyclin Dependent Kinase (CDK)N2a
Brief Title: Cyclin Dependent Kinase (CDK)4/6 Inhibitor, PD0332991 in Advanced Non-small Cell Lung Cancer NSCLC.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD0332991
Record Dates: First submitted 2011-02-01; First posted 2011-02-07 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Advanced stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD0332991 (Experimental): PD0332991 125 mg PO days 1 - 21
  Interventions: Drug: PD0332991

INTERVENTIONS:
Drug: PD0332991 — PD0332991 125 mg PO days 1 - 21
  Other Names: Palbociclib

SUMMARY:
The purpose of this study is to determine the efficacy and the toxicities of the study drug PD0332991 in the treatment of patients with Stage IV non-small cell lung cancer with wildtype retinoblastoma protein (RB) and inactivated cyclin dependent kinase (CDK) N2A in the tumor.

DETAILED DESCRIPTION:
The oral drug PD0332991 is a highly selective reversible inhibitor of cyclin-dependent kinases 4 & 6 that is being studied for use in the treatment of advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven non small cell lung cancer
* Stage IV (M1a or M1b) disease. Patients may also have recurrence of early-stage disease or locally advanced disease with the presence of new distant metastases.
* Cyclin dependent kinase (CDK)N2a (p16) protein absent or expressed at a low level in tumor biopsy specimen
* Failed or intolerant of at least one prior systemic chemotherapy regimen (there is no maximum number of prior chemotherapy regimens)
* Eastern cooperative oncology group (ECOG) performance status 0-2
* Age >18 years.
* Adequate organ and bone marrow function
* Measurable disease by standard RECIST v1.1 criteria
* Life expectancy of greater than 3 months

Exclusion Criteria:

* Inability to understand or sign the informed consent document
* Inability or unwillingness to take oral medications
* No available tissue specimen for p16 analysis
* Chemotherapy or radiotherapy within 3 weeks prior to beginning the study drug
* Other investigational agents within 4 weeks prior to beginning the study drug
* All side effects from previous chemotherapy, radiotherapy or investigational agents not resolved, returned to baseline or returned to Grade 1 toxicity (exceptions are grade 2 alopecia and grade 2 peripheral neuropathy)
* Major surgery within 4 weeks prior to beginning the study drug
* Surgical scar from previous surgery not healed prior to beginning the study drug
* High-dose or chronic steroid use
* High-dose statins within 7 days
* History of rhabdomyolysis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes, stroke or myocardial infarction within 3 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Baseline corrected QT interval (QTc) >470ms
* Pre-existing clinically significant cardiac, hepatic or renal dysfunction at the discretion of the treating physician
* Untreated or uncontrolled (symptomatic or asymptomatic) brain metastases
* Leptomeningeal carcinomatosis
* Inability or unwillingness to use contraception during the treatment period by patients with reproductive potential.
* Pregnant or breastfeeding women
* HIV-positive patients on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Gopalan, MD, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health Cancer Center, Gainesville, Florida
  - H. Lee Moffitt Cancer and Research Institute, Tampa, Florida

REFERENCES:
- See also: UF Health Cancer Center — http://cancer.ufl.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PD0332991
Started | 19
Completed | 14
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | PD0332991
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response by Direct RECIST Measurement
Description: Response is a decrease in the sum of the longest diameters of the target lesions by more than 30% compared to the baseline.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | PD0332991
Number analyzed (Participants) | 16
participants | 0

2. Secondary Outcome: Overall Survival
Description: Median overall survival
Time Frame: 14 months
Measure: Median (Standard Error); unit: weeks
Arm/Group | PD0332991
Number analyzed (Participants) | 14
weeks | 20.3 (1.7)

3. Secondary Outcome: Progression-free Survival
Description: Median progression-free survival.
Time Frame: 12 months
Measure: Median (Standard Error); unit: Weeks
Arm/Group | PD0332991
Number analyzed (Participants) | 16
Weeks | 8 (0.7)

4. Secondary Outcome: Plasma Levels
Description: Plasma levels of p16, phosphorylated RB and cyclin d1 in blood.
Time Frame: 6 months
Population: 4 of the 16 samples were tested by protein immunoblot (Western blot), and due to the test not being sensitive enough to detect p16, phosphorylated RB or cyclin D1 protein bands in any of the samples, the decision was made not to purse this testing any further.
Measure: Number; unit: Arbitrary Units
Arm/Group | PD0332991
Number analyzed (Participants) | 4
Arbitrary Units | NA — 4 of the 16 samples were tested by Western blot, and due to the test not being sensitive enough to detect p16, phosphorylated RB or cyclin D1 protein bands in any of the samples, the decision was made not to pursue this testing any further.

5. Secondary Outcome: Grade of Study Drug Toxicity
Description: The number of all toxicities and grades 3 and 4 (per CTCAE v3.0) toxicities that occured during the administration of the drug and during the follow up period.
Time Frame: 24 months
Measure: Number; unit: Events
Arm/Group | PD0332991
Number analyzed (Participants) | 16
Events
  Grade 3 and 4 Toxicities | 9
  All Toxicities (Grades 1 - 5) | 86

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the Informed Consent Form through 30 days after the last dose of study drug (approximately 20 weeks).
Description: All adverse events were assessed using the results of routine bloodwork, imaging or by a qualified healthcare provider.
Arm/Group | PD0332991
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD0332991 (N=19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD0332991 (N=19)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 9 (13)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Chills (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify: Body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify: Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10)
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 (7)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (5)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus (General disorders) | 1 (2)
Psychiatric disorders - Other, specify: Mood changes (Psychiatric disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8)
Watering eyes (Eye disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No